CLINICAL TRIAL: NCT06029569
Title: Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of Rapamycin Coated Balloon Dilation Catheter in the Treatment of Dialysis Pathway Stenosis or Blockage in Hemodialysis Patients
Brief Title: Rapamycin Coated Balloon Dilation Catheter for Arteriovenous Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Bomaian Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMA-AVF-DCB
Record Dates: First submitted 2023-08-24; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapamycin coated balloon dilation catheter for arteriovenous fistula (Experimental): Experimental group rapamycin balloon therapy for autologous arteriovenous fistulas with stenosis or occlusion
  Interventions: Procedure: Rapamycin drug balloon angioplasty; Procedure: Paclitaxel drug balloon angioplasty
- Paclitaxel release high-pressure shunt balloon dilation catheter (Sham Comparator): Strict or occluded autologous arteriovenous fistula treated with paclitaxel balloon therapy in the control group
  Interventions: Procedure: Rapamycin drug balloon angioplasty; Procedure: Paclitaxel drug balloon angioplasty

INTERVENTIONS:
Procedure: Rapamycin drug balloon angioplasty — Rapamycin drug balloon treatment for stenosis or blockage of the dialysis pathway in autologous arteriovenous fistula.
Procedure: Paclitaxel drug balloon angioplasty — Paclitaxel drug balloon therapy for stenosis or blockage of the dialysis pathway of autologous arteriovenous fistula.

SUMMARY:
Verify the effectiveness and safety of rapamycin coated balloon dilation catheter for the treatment of dialysis pathway stenosis or blockage lesions.

DETAILED DESCRIPTION:
To verify the effectiveness and safety of the Rapamycin coated arteriovenous fistula balloon dilation catheter developed and produced by Shanghai Bomaian Medical Technology Co., Ltd. in the treatment of stenosis or blockage of the dialysis pathway of autologous arteriovenous fistula in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. AVF has been established, with mature development and at least one successful completion of hemodialysis；
2. AVF has significant hemodynamic abnormalities；

exclusion criteria

1. The target lesion has undergone intervention treatment within 30 days；
2. An intravascular stent has been placed at any location along the vascular pathway；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
6-month target lesion primary patency rate | 6months
  Primary patency is defined as puncture dialysis that can be used to meet the requirements of the dialysis prescription without intervention treatment after the target lesion surgery.

SECONDARY OUTCOMES:
Device success rate | The day of operation.
  The treatment device can be successfully transported, expanded, and withdrawn without any defects such as balloon rupture or loss of device integrity or design performance when expanded without exceeding the rated burst pressure.
Surgical success rate | 7Days
  The residual stenosis of the target lesion is ≤ 30%, and there are no adverse events related to the target dialysis pathway related to medical devices within 7 days after surgery/before discharge.
Clinical success rate | 1year
  After the surgery, at least one puncture dialysis that meets the requirements of the dialysis prescription has been completed and no target pathway dysfunction has occurred before.

IPD SHARING:
Plan to Share IPD: No